CLINICAL TRIAL: NCT06923605
Title: The Efficacy of Erythropoietin Oral Gel Versus Erythropoietin Mouthwash in the Management of Recurrent Aphthous Stomatitis: A Randomized Controlled Clinical Study With Biochemical Analysis
Brief Title: The Efficacy of Erythropoietin Oral Gel Versus Erythropoietin Mouthwash in the Management of Recurrent Aphthous Stomatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mai Talaat Mohamed, lecturrer assistant, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAsu-Rec ID032209
Record Dates: First submitted 2025-03-11; First posted 2025-04-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Erythropoietin; IL-2; Recurrent aphthous stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Erythropoietin/oral gel (Experimental): topical erythropoietin oral gel 4 times daily for 1 week
  Interventions: Drug: Epoetin 4000
- placebo (Experimental): isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl) 4 times daily
  Interventions: Other: Placebo
- Erythropoietin/mouthwash (Experimental): Erythropoietin mouthwash 4 times daily for 1 week
  Interventions: Drug: Epoetin 4000

INTERVENTIONS:
Drug: Epoetin 4000 — Erythropoietin hormone
  Arms: Erythropoietin/mouthwash; Erythropoietin/oral gel
Other: Placebo — isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl) 4 times daily
  Arms: placebo

SUMMARY:
Erythropoietin (EPO) exerts anti-inflammatory effects by inhibiting NF- kappa B-dependent formation of pro-inflammatory cytokines, thus it reduces local and circulating levels of these disease (recurrent aphthous stomatitis RAS) related cytokines. So, it is considered as a potent anti-inflammatory cytokine in inflammatory disorders and infectious disease. It also accelerates wound-healing and decreases the extent of apoptosis and the areas of the open wound. this drug seems to be a promising therapeutic option in oral lesions. the effectiveness of EPO oral gel and EPO mouth wash were compared on patients with recurrent aphthous stomatitis and investigated therapeutic mechanism by examining treatment effect on expression of IL-2 IN RAS.

DETAILED DESCRIPTION:
Sixty patients with recurrent aphthous stomatitis were randomly assigned into three equal groups to receive topical Erythropoietin oral gel four times per day (after meals and at bedtime) (Group I).

Erythropoietin mouthwash 4 times per day (after meals and at bedtime) (Group II), and placebo isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl) (Group III).

All patients were followed up four 1 week, photographs were taken at the beginning and end of the treatment.

patients were assessed using pain visual analogue scale (PVAS), clinical assessments for the size of the ulcers and rate of their recurrence.

pretreatment and post treatment salivary samples were taken to detect the expression and levels of salivary IL-2.

ELIGIBILITY:
Inclusion Criteria:

* All patients should be free from any systemic disease or Behcet syndrome.
* Patients ≥18 years of age, male or female are eligible.
* Oral pain score of 4 or higher on a scale of 0-10 with 0 representing no pain in the presence of oral ulceration.
* Patient has only aphthous ulcer and It should had not been passed more than 4 days from beginning of their ulcer.

Exclusion Criteria:

* • Patients with poor oral hygiene or not willing to perform oral hygiene measures.

  * Smoking and alcohol use.
  * Pregnant and lactating females
  * Patients with history of any topical or systemic medication or steroid therapy 1 month prior to the investigation.
  * The vulnerable group; prisoners, mentally or physically disabled patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Pain visual analogue scale (P-VAS) | Reduction from baseline and after 1 week of treatment
  The pain VAS consisted of a 10-cm horizontal line marked 0-10 (0 no pain, 10 most severe pain experienced). Patients marked the scale at each visit, and the all P-VAS were included on one sheet of paper allowing the patient to think in terms of change instead of absolutes. The P-VAS was then scored by measuring from the patient's mark to the beginning of the scale in cm.

SECONDARY OUTCOMES:
Size of the ulcer | change from baseline and after 1 week of treatment
  The score corresponds to the average diameter of the ulcers in millimeters, that is, a patient having ulcers of average size of 5 mm would score 5. Patients indicated the average size of their ulcers on a diagram of different diameter circles. The maximum score was 20 to accommodate the small number of RAS cases in which ulcers are on average more than 10 mm in diameter.

OTHER OUTCOMES:
Biochemical analysis | From baseline and after 1 week of treatment
  Salivary IL-2 was detected by an Enzyme-Linked Immunosorbent Assay (ELISA). This sandwich kit is for the accurate quantitative detection of Human Interleukin 2 (also known as IL-2) in serum, plasma, cell culture supernates, Ascites, tissue homogenates or other biological fluids.

CONTACTS AND LOCATIONS:
Overall Officials: Mai T. assistant lecturer Mai T. Elgendi, Assistant lecturer, Study Director — Faculty of oral medicine- Future University in Egypt
Locations (1):
- Future university in Egypt, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the age and number of the participants
Supporting Information: Study Protocol, ICF
Time Frame: will be available in September 2025
Access Criteria: other researchers in oral medicine will be able to access, when the experiment is published internationally
URL: http://clinicaltrials.gov

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov